CLINICAL TRIAL: NCT01058785
Title: Phase II Study of Lucanix™ (TGF-beta2 Antisense Gene Modified Allogeneic Tumor Cell Vaccine) in Patients With Stages II-IV Non-Small Cell Lung Cancer
Brief Title: Phase II Study of Lucanix™ in Patients With Stages II-IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaRx Corporation (Industry)
Responsible Party: Habib Fakhrai, Ph.D., NovaRx Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-IND 8868
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-01

CONDITIONS: Lung Neoplasm; Carcinoma, Bronchogenic
Keywords: Gene therapy; Flow cytometry; Immunoenzyme technique; Laboratory biomarker analysis; Tumor cell-derivative vaccine therapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Bronchogenic | interventions — belagenpumatucel L

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lucanix (Experimental): Patients will receive injections of Lucanix for each dose cohort.
  Interventions: Biological: Lucanix

INTERVENTIONS:
Biological: Lucanix — Monthly intradermal injections of four irradiated allogeneic TGF-beta2 antisense gene modified NSCLC cell lines. Patients are randomized to receive either 12,500,000, 25,000,000 or 50,000,000 cells per injection for up to 16 injections.
  Other Names: belagenpumatucel-L

SUMMARY:
In this Phase II clinical trial the investigators will use four human non-small cell lung cancer cell lines that have been previously established in tissue culture laboratory. The investigators will gene modify these tumor cells in the laboratory to block their TGF-beta secretion. The investigators will inject the genetically engineered cells as vaccines in patients with stages II to IV non-small cell lung cancer. Our rationale for using other people's tumor cells is that lung tumor cell lines belonging to different people have been shown to share common characteristics that are recognized by non-self immune systems.

DETAILED DESCRIPTION:
This will be a 2-stage, open-label, three-arm, Phase II study. It is designed to evaluate the efficacy of immunization with increasing doses of an allogeneic tumor cell vaccine, Lucanix™, in patients with non-curable NSCLC. Patients will be followed for clinical response, immunogenicity and safety.

Eligible patients will receive 4 monthly intradermal injections with a cell cocktail comprised of equal numbers of four irradiated allogeneic TGF-beta2 antisense gene modified NSCLC cell lines. Patients will be randomized to one of the three study cohorts. Patients will receive 12,500,000, 25,000,000, 50,000,000 gene modified cells respectively. Treated patients will be evaluated four months after they enter therapy. Patients that respond to therapy will receive an additional four to twelve injections to evaluate whether their response to therapy can be amplified. Response, time to tumor progression, and tumor free survival will be monitored in patients and compared with historical controls and patients receiving other forms of therapy. Patients will be monitored and evaluated according to standard evaluation criteria of no response, stable disease, partial response and complete response.

PRIMARY OBJECTIVE

-Evaluate the ability of increasing doses of Lucanix™, a gene-modified tumor cell vaccine, to induce tumor response in patients with non-curable NSCLC

SECONDARY OBJECTIVES

* Evaluate the ability of the Lucanix™ vaccination regimen to induce an immune response (cellular and humoral)
* Estimate the response duration for the Lucanix™ regimen
* Evaluate the effects of repeated inoculations on immune infiltrates
* Evaluate the safety of the Lucanix™ regimen

INCLUSION CRITERIA

* Signed informed consent
* 18 years
* Histologically confirmed non-curable NSCLC with an estimated total tumor burden volume of less than or equal to 125 cc, confirmed to be stage II, III, or IV.
* Must have completed or refused conventional therapy
* Performance status (ECOG) less than 2.
* Absolute granulocyte count greater than or equal to 1,500/mm3
* Platelet count greater than or equal to 100,000/mm3
* Total Bilirubin less then or equal to 2 mg/dL
* AST and ALT less than or equal to 2x Upper Limit of Normal
* Creatinine less than or equal to 1.5 mg/dL

EXCLUSION CRITERIA

* Concurrent systemic steroids greater than 2 mg prednisone/day
* Prior splenectomy
* Any surgery involving general anesthesia, chemotherapy, radiotherapy, steroid therapy or immunotherapy less than 4 weeks of study entry
* Brain metastases or meningeal lymphomatosis unless treated and stable for greater than or equal to 2 months
* Known HIV positive
* Serious non-malignant disease (e.g., congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections), or other conditions which, in the opinion of the investigator would compromise protocol objectives.
* Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for greater than or equal to 2 years
* Treatment with an investigational drug within 30 days prior to study entry
* History of psychiatric disorder that would impede adherence to protocol
* Pregnant or nursing women or refusal to practice contraception if of reproductive potential

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years
* Histologically confirmed non-curable NSCLC with an estimated total tumor burden volume of less than or equal to 125 cc, confirmed to be stage II, III, or IV.
* Must have completed or refused conventional therapy
* Performance status (ECOG) less than 2.
* Absolute granulocyte count greater than or equal to 1,500/mm3
* Platelet count greater than or equal to 100,000/mm3
* Total Bilirubin less than or equal to 2 mg/dL
* AST and ALT less than or equal to 2x Upper Limit of Normal
* Creatinine less than or equal to 1.5 mg/Dl

Exclusion Criteria:

* Concurrent systemic steroids greater than 2 mg prednisone/day
* Prior splenectomy
* Any surgery involving general anesthesia, chemotherapy, radiotherapy, steroid therapy or immunotherapy less than 4 weeks of study entry
* Brain metastases or meningeal lymphomatosis unless treated and stable for ≥ 2 months
* Known HIV positive
* Serious non-malignant disease (e.g., congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections), or other conditions which, in the opinion of the investigator would compromise protocol objectives.
* Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for greater than or equal to 2 years
* Treatment with an investigational drug within 30 days prior to study entry
* History of psychiatric disorder that would impede adherence to protocol
* Pregnant or nursing women or refusal to practice contraception if of reproductive potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the ability of increasing doses of Lucanix™, a gene-modified tumor cell vaccine, to induce tumor response in patients with non-curable NSCLC | Week 16, quarterly during treatment and first year of post-intervention follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Habib Fakhrai, PhD, Study Director — NovaRx Corporation
Locations (3):
- United States (3):
  - Hoag Cancer Center, Newport Beach, California
  - Jayne Gurtler MD, Laura Brinz MD, Angelo Russo MD, and Janet Burroff MD APM, Metairie, Louisiana
  - Mary Crowley Medical Research Center, Dallas, Texas

REFERENCES:
- [Background] Fakhrai H, Mantil JC, Liu L, Nicholson GL, Murphy-Satter CS, Ruppert J, Shawler DL. Phase I clinical trial of a TGF-beta antisense-modified tumor cell vaccine in patients with advanced glioma. Cancer Gene Ther. 2006 Dec;13(12):1052-60. doi: 10.1038/sj.cgt.7700975. Epub 2006 Jul 7. PMID 16826191
- [Result] Nemunaitis J, Dillman RO, Schwarzenberger PO, Senzer N, Cunningham C, Cutler J, Tong A, Kumar P, Pappen B, Hamilton C, DeVol E, Maples PB, Liu L, Chamberlin T, Shawler DL, Fakhrai H. Phase II study of belagenpumatucel-L, a transforming growth factor beta-2 antisense gene-modified allogeneic tumor cell vaccine in non-small-cell lung cancer. J Clin Oncol. 2006 Oct 10;24(29):4721-30. doi: 10.1200/JCO.2005.05.5335. Epub 2006 Sep 11. PMID 16966690
- See also: Clinical trial information — http://www.novarx.com/